CLINICAL TRIAL: NCT05647356
Title: The RolE oF Androgen Excess in MUscle Energy MetaboLism in Women With PolyCystic Ovary Syndrome (REFUEL PCOS) Study 2
Acronym: REFUEL PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University of Birmingham (Other); University of Liverpool (Other); University of Oxford (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Michael W, Professor, Royal College of Surgeons, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22/52
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Polycystic Ovary Syndrome; Androgen Excess; Metabolic Disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Metabolic Diseases | interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bicalutamide (Experimental): Adult females with polycystic ovary syndrome (PCOS) and evidence of clinical or biochemical androgen excess will be recruited.
  Interventions: Drug: Bicalutamide 50 mg

INTERVENTIONS:
Drug: Bicalutamide 50 mg — Bicalutamide at a dose of 50mg once daily for 28 days.

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 10% of all women, and it usually co-exists with high levels of sex hormones called androgens, such as testosterone. Women with PCOS are at increased risk of metabolic complications such as diabetes, non-alcoholic fatty liver disease, high blood pressure and heart disease. However, very little is understood about how androgen excess may drive the metabolic complications observed in women with PCOS.

Skeletal muscle is an important site of energy metabolism; increasingly, it is suspected that skeletal muscle energy balance is adversely impacted by androgens, thereby driving metabolic complications. To take this theory forward, we want to investigate the effects of androgens on muscle energy metabolism. We will perform detailed metabolic testing (including blood tests and muscle biopsies) in women with PCOS before and after taking tablets that block the action of testosterone for 28 days. In addition, we will be using a gold standard technique to see how women with PCOS metabolise fat and other nutrients by measuring markers in blood and breath samples after a breakfast test meal. This clinical research will increase our understanding of the complex relationships between hormonal abnormalities and metabolic disease in women with PCOS.

DETAILED DESCRIPTION:
Background:

Polycystic ovary syndrome (PCOS) is a lifelong metabolic disorder affecting 10-13% of all women and is associated with major healthcare and economic burden, estimated at $8 billion annually the US in 2020. Traditionally considered a reproductive disorder only, it is now increasingly clear that PCOS is associated with severe metabolic health consequences across the entire life course of women. There is a two-fold increased risk of type 2 diabetes mellitus (T2DM), nonalcoholic fatty liver disease, and emerging evidence of increased cardiovascular disease (CVD) incidence. There are no disease-specific therapies to mitigate or treat metabolic risk in women with PCOS. This is consistently highlighted as the priority concern amongst PCOS patient advocacy groups.

Androgen excess is a cardinal feature of PCOS, and circulating androgen burden is closely correlated with metabolic complications. In women with PCOS, the risk of developing metabolic dysfunction is above that conferred by simple obesity, suggesting that androgen excess is a key player; however, a distinct mechanistic role for androgens in this process remains to be elucidated. Androgen excess is associated with metabolically deleterious visceral fat accumulation and circulating testosterone levels correlate directly with the risk of T2DM and NAFLD. Muscle is a critical metabolic target tissue that plays a central role in energy metabolism through processes such as glucose uptake and oxidation, as well as oxidation of fatty acids to generate ATP in the mitochondria. Recent mechanistic data have shown that androgen excess is associated with changes in the transcriptional profile of skeletal muscle genes linked with metabolism and energy balance. Therefore, skeletal muscle is likely to represent an important site of crosstalk between androgen excess, disturbances in energy metabolism and risk of metabolic disease in PCOS.

Defective skeletal muscle glucose uptake is a key early step in the pathogenesis of insulin resistance in PCOS, and an early predictor of progression to overt type 2 diabetes mellitus. Impaired mitochondrial oxidation of free fatty acids in skeletal muscle and other disturbances in skeletal muscle mitochondrial function, such as oxidative phosphorylation, are increasingly implicated in the pathogenesis of metabolic disease such as T2DM. Abnormalities in skeletal muscle mitochondrial function have also been identified in small-scale studies in women with PCOS, and were associated with impaired fatty acid oxidation, weight gain and an increased risk of diabetes.

We hypothesise that androgen-mediated disturbances in skeletal muscle energy balance play a major role in the pathogenesis of metabolic disease in women with PCOS.

Study description:

We propose to test our hypothesis utilising state-of-the-art metabolic phenotyping tools in two study visits. We will examine systemic fatty acid oxidation, muscle proteomics and targeted and non-targeted metabolomics in women with PCOS before and after pharmacological androgen receptor blocade. In addition, a subset of ex vivo muscle biopsies will undergo in vitro experiments to measure skeletal muscle mitochondrial morphology and function.

After study visit 1, all recruited participants will receive 50mg of an oral androgen receptor antagonist (bicalutamide), resulting in pharmacological AR blockade, before undertaking an identical study visit for repeat assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women with a confirmed diagnosis of polycystic ovary syndrome with androgen excess on clinical or biochemical grounds
* BMI 20-40kg/m2
* Age range 18-40 years
* Ability to provide informed consent
* Negative pregnancy test at screening
* Effective method of contraception (will sign a pregnancy waiver)

Exclusion Criteria:

* A confirmed diagnosis of diabetes
* Current or recent (<3 months) use of weight loss medications
* Current or recent use of oral contraceptive pill or hormone replacement therapy (within last 3-months)
* Blood haemoglobin <11.0g/dL
* History of alcoholism or a greater than recommended alcohol intake (recommendations > 21 units on average per week for men and > 14 units on average per week for women)
* Haemorrhagic disorders
* Treatment with anticoagulant agents
* Other co-morbidities that in the view of the investigators may affect data collection
* Any medical condition in the opinion of the investigator that might impact upon safety or validity of the results
* Pregnancy or breastfeeding at the time of planned recruitment
* A diagnosis of PCOS according to Rotterdam criteria where the patient does not have clinical or biochemical evidence of androgen excess
* History of significant renal (eGFR<30) or hepatic impairment (AST or ALT >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
* Any other significant disease or disorder that, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational medicinal product in the 12 weeks preceding the planned recruitment
* Glucocorticoid use via any route within the last three months
* Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment
* Use of oral or transdermal hormonal contraception in the three months preceding the planned recruitment
* Use of contraceptive implants in the twelve months preceding the planned recruitment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with a confirmed diagnosis of polycystic ovary syndrome with androgen excess on clinical or biochemical grounds
Enrollment: 16 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To examine the impact of androgen receptor blockade (AR) on systemic and muscle-specific energy metabolism in women with PCOS and androgen excess | 2.5 years
  Change in whole body fatty acid oxidation on stable isotope breath after 28 days of androgen receptor (AR) blockade compared to baseline

SECONDARY OUTCOMES:
To determine the relationship between androgen excess and serum/muscle non-targeted metabolomics | 2.5 years
  Changes in metabolomic pathways relating to energy balance and mitochondrial function in serum and muscle after AR blockade
To determine the impact of androgen receptor blockade on skeletal muscle mitochondrial morphology and function ex vivo | 2.5 years
  Changes in mitochondrial morphology ex vivo post AR blockade
To determine the impact of androgen receptor blockade on skeletal muscle mitochondrial morphology and function ex vivo | 2.5
  Differences in mitochondrial oxygen consumption and oxidative phosphorylation using Seahorse technology pre and post AR blockade

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Collage Of Surgeons, Dublin, Ireland